CLINICAL TRIAL: NCT07171320
Title: Comparing the Efficacy and Safety of Pregabalin Monotherapy With Pregabalin Combined Other Neuromodulatory Drugs (Desvenlafaxine) in the Treatment of Fibromyalgia: A Multicenter Clinical Study
Brief Title: The Efficacy and Safety of Pregabalin Combined With Desvenlafaxine in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Jiujiang University Affiliated Hospital (Other Government)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-217-03-04
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Pregabalin; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin; Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin monotherapy group (Active Comparator)
  Interventions: Drug: Pregabalin
- Pregabalin with desvenlafaxine group (Experimental)
  Interventions: Drug: Pregabalin with desvenlafaxine

INTERVENTIONS:
Drug: Pregabalin — In the pregabalin monotherapy group, pregabalin will be initiated at 150 mg daily, divided into 2 or 3 doses per day, and increased to 300 mg per day after 3 to 7 days, subsequent increases of 150 mg daily may occur every 3 to 7 days, based on individual patient response and tolerability, with a maximum dose of 600 mg daily.
  Arms: Pregabalin monotherapy group
Drug: Pregabalin with desvenlafaxine — In the pregabalin with desvenlafaxine group, the dose titration of pregabalin is identical with pregabalin monotherapy group. Desvenlafaxine will be administered at 50 mg daily with breakfast initially. If the initial dose is well-tolerated, the dose could be further escalated by 50 mg per day after 3 days, up to a maximum of 400 mg per day after 7 days. With each dose increase, AEs will be assessed and categorized as mild, moderate, or severe. If participants tolerate the current dose for 2 to 3 days, it will be maintained, with the expectation that tolerance to AEs will develop. If AEs become intolerable, the dose will be decreased back to the previous dose, which was defined as the maximum tolerated dose. In the combination group, dose titration of both pregabalin and desvenlafaxine will be conducted simultaneously. If AEs occur, the next dose regimen should be determined in consultation with a clinical physician.
  Arms: Pregabalin with desvenlafaxine group

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread pain, fatigue, and emotional disorders. Its onset is related to factors such as central sensitization and imbalance of neurotransmitters. The current mainstream treatments include pregabalin, but the efficacy of pregabalin is limited, with only 25%-40% pain relief rate, and adverse reactions are common. Selective serotonin and norepinephrine reuptake inhibitors (SNRIs), such as duloxetine and venlafaxine, have demonstrated efficacy in FM by modulating pain pathways through increased serotonin and norepinephrine availability. Desvenlafaxine, the third SNRI, was found with lower adverse effects compared with duloxetine and venlafaxine. We hypothesize that the combination of pregabalin with desvenlafaxine may offer greater pain relief compared pregabalin monotherapy, without a significant increase in adverse effects for patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FM according to the 2016 Revisions to the 2010/2011 FM diagnostic criteria;
* Aged 18 years or older;
* Experiencing moderate to severe FM that have not been effectively alleviated by non-pharmacological treatments and has not received currently recommended pharmacological treatment for FM;
* Numeric rating scale (NRS) score ≥ 4 at baseline;
* Aspartate aminotransferase and alanine aminotransferase levels less than twice the upper limit of normal;
* Estimated glomerular filtration rate of 30 mL/min per 1.73 m2 or higher;
* Willing to sign the informed consent form and possessing sufficient cognitive and language abilities to comply with all the study requirements.

Exclusion criteria

* History of hypersensitivity to pregabalin, desvenlafaxine or any of its excipients;
* History of epilepsy, or depression requiring antidepressant medications;
* Pregnancy or breastfeeding;
* Presence of serious systemic diseases, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac dysfunction;
* With acute or chronic pain conditions other than FM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The average pain intensity | at the 4-weeks
  The average pain intensity over the past 24 hours, rated each morning upon awakening and averaged over 7 days at the 4 weeks. This will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
The worst pain intensity | At the weeks 1, 2, 4, and 8
  The worst pain intensity over the past 24 hours, rated each morning upon awakening and averaged over 7 days. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
The proportion of patients achieving pain reduction | At the weeks 1, 2, 4, and 8
  The proportion of patients achieving a ≥ 50% and ≥ 30% reduction in mean baseline pain intensity. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
The Revised FM Impact Questionnaire | At the weeks 1, 2, 4, and 8
  The Revised FM Impact Questionnaire assesses the severity of FM symptoms and their impact on daily functioning. It evaluates three linked domains: function, overall impact, and symptoms, using a 0 to10 NRS. The total score ranges from 0 to 100, with higher scores indicating greater disease burden.
The Brief Pain Inventory (BPI) severity (BPI-S) and interfere (BPI-I) subscales | At the weeks 1, 2, 4, and 8
  BPI-S accesses pain intensity over the past 24 hours, calculated as the average of items 3 to 6 on the BPI, scored using a 0 to 10 NRS. In the NRS scale, 0 indicates no pain, while 10 represents the worst pain imaginable. The total score ranges from 0 to 40, with higher scores indicating greater pain severity. BPI-I evaluates the degree to which pain interferes with daily activities, including general activity, mood, mobility work, relationships, sleep, and pleasure. This subscale comprises 7 items, each scored from 0 (no interference) to 10 (complete interference), with a total score ranging from 0 to 70.
The short-form 36 Health Survey (SF-36) | At the weeks 1, 2, 4, and 8
  The SF-36 assesses health-related quality of life, capturing preferences across various health states. It assesses 8 dimensions: physical functioning, physical role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional role limitations due to emotional problems, and mental health. Scores range from 0 to 100 for each dimension, with higher scores indicating better health status.
The Medical Outcomes Study Sleep Scale (MOS) | At the weeks 1, 2, 4, and 8
  The MOS is a questionnaire comprising 12 items that assess various aspects of sleep using a 6-point ordinal scale (1 indicating permanence and 6 indicating absence).
The Beck Depression Inventory-Ⅱ (BD-Ⅱ) | At the weeks 1, 2, 4, and 8
  The BD-Ⅱ evaluates the severity of depressive symptoms using a 4-point scale from 0 to 3, where 0 indicates no symptom and 3 indicates severe symptomatology. It comprises 21 items, the total score ranging from 0 to 63.
Adverse Events | Through study completion, an average of 8 weeks
  The incidence and proportion of adverse events will be recorded and categorized as mild, moderate, severe, or life-threatening. AEs are defined as events that arise during treatment, were absent before treatment, or worsen relative to the pretreatment state.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Mathieson S, Lin C-WC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020;369:m1315. doi: 10.1136/bmj.m1315 — https://pubmed.ncbi.nlm.nih.gov/32345589/
- See also: Domon Y, Arakawa N, Inoue T, Matsuda F, Takahashi M, Yamamura N, et al. Binding Characteristics and Analgesic Effects of Mirogabalin, a Novel Ligand for the α2δ Subunit of Voltage-Gated Calcium Channels. J Pharmacol Exp Ther. 2018;365(3):573-82. doi: 10. — https://pubmed.ncbi.nlm.nih.gov/29563324/
- See also: Migliorini F, Maffulli N, Eschweiler J, Baroncini A, Bell A, Colarossi G. Duloxetine for fibromyalgia syndrome: a systematic review and meta-analysis. J Orthop Surg Res. 2023;18(1):504. doi: 10.1186/s13018-023-03995-z. — https://pubmed.ncbi.nlm.nih.gov/37461044/
- See also: Gilron I, Chaparro LE, Tu D, Holden RR, Milev R, Towheed T, et al. Combination of pregabalin with duloxetine for fibromyalgia: a randomized controlled trial. Pain. 2016;157(7):1532-40. doi: 10.1097/j.pain.0000000000000558. — https://pubmed.ncbi.nlm.nih.gov/26982602/